CLINICAL TRIAL: NCT00026091
Title: Phase II Trial of Fenretinide (NSC 374551) in Recurrent Ovarian Cancer and Primary Peritoneal Carcinoma
Brief Title: Fenretinide in Treating Patients With Recurrent or Metastatic Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00457; PHII-25; N01CM17101 (NIH); CDR0000068985 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Fenretinide

ARMS (1):
- Treatment (fenretinide) (Experimental): Patients receive oral fenretinide twice daily on days 1-7. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fenretinide; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: fenretinide — Given orally
  Other Names: fenretinimide; McN-R-1967
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of fenretinide in treating patients who have recurrent or metastatic ovarian epithelial or primary peritoneal cancer. Drugs used in chemotherapy, such as fenretinide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of fenretinide (4-HPR) in patients with recurrent ovarian cancer or primary peritoneal carcinoma.

II. To assess the toxicity of this agent in this patient population. III. To evaluate molecular changes in normal and tumor cells induced by 4-HPR by studying: (a) the analysis of ceramide and glucosyleceramide levels before and after therapy, (b) intracellular levels of 4-HPR and 4-MPR, and (c) determinants of apoptosis (p53, p21, bcl-2, bax and terminal deoxynucleotidyl transferase [TdT] assay) in baseline tumor specimens, serial serum and tumor biopsy specimens where available, and surrogate in-vitro studies.

IV. To evaluate the pharmacokinetics of fenretinide. V. To further investigate the antiangiogenesis effects of fenretinide in in-vitro assays using ovarian cancer cell lines and in vascular growth factor (VEGF, TGFb) plasma levels in patients.

OUTLINE:

Patients receive oral fenretinide twice daily on days 1-7. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed recurrent or metastatic epithelial ovarian cancer or primary peritoneal carcinoma
* Unidimensionally measurable disease; indicator lesions must not have been irradiated unless they have grown following radiation therapy
* SWOG performance status 0-2
* Patients must have received a platinum and paclitaxel containing regimen
* Patients are allowed to receive =< 2 prior chemotherapy regimens for recurrent disease; patients who are rechallenged with the same chemotherapy regimen are considered to have had that regimen only once
* Projected life expectancy must be at least 3 months
* Signed informed consent
* Absolute neutrophil count >= 1500/ul
* Platelet count >= 100,000 ul
* Bilirubin =< 2 times the institutional limit of normal
* ALT or AST =< 3 times the upper limit of normal
* Measured or calculated creatinine clearance >= 60 ml/min
* Fasting triglycerides =< 1 time the upper limit of normal; triglycerides may be "normalized" prior to study entry with use of an antilipemic agent (atorvastatin, fenofibrate)
* Patients must have recovered from acute toxicities from surgery, radiation or chemotherapy; at least 3 weeks will have elapsed since any prior therapy directed at the malignant tumor
* Patients of childbearing potential must agree to use an approved method of birth control

Exclusion Criteria:

* Prior fenretinide is not allowed; prior 13-cis, 9-cis or all-transretinoic acid are allowed
* Patients with a second malignancy within the last 5 years are not allowed, except for those with non-melanomatous skin cancer and carcinoma-in-situ of the cervix; all prior invasive malignancies must be in complete remission
* The use of concomitant antioxidants, such as vitamin C or E, is not allowed
* Patients with concurrent medical, psychological or social conditions of such severity that the investigator deems it unwise to enter the patient on protocol
* Untreated or symptomatic brain metastases
* Pregnant or nursing women

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-09; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Response rate (CR or PR) | Up to 9 years
  Associated exact 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Time to treatment failure | up to 9 years
  Estimated using the product-limit method of Kaplan and Meier.
Duration of response | From the time measurement criteria met for CR/PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 9 years
  Estimated using the product-limit method of Kaplan and Meier.
Overall survival | From first day of treatment to time of death due to any cause, assessed up to 9 years
  Estimated using the product-limit method of Kaplan and Meier.
Toxicity | Up to 9 years after completion of treatment
  Tables will be constructed to summarize the observed incidence by severity and type of toxicity.
Pharmacokinetics of fenretinide | Baseline. day 1, 4 and 7 of courses 1, day 1 of courses 2, 5, and 9, day 7 of courses 4 and 8
  Summarized with simple summary statistics: means or medians, ranges, and standard deviations (if numbers and distribution permit).
Molecular change | Baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States